CLINICAL TRIAL: NCT02589951
Title: Missed Serious Medical Illness in Psychiatric Patients Seen in an Academic Emergency Department
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: REB 107073
Record Dates: First submitted 2015-10-26; First posted 2015-10-28 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Psychiatric Patients, Serious Medical Illness

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: admission to non-psychiatric service

SUMMARY:
The purpose of this study is to determine the prevalence, etiology, and timing of missed Serious Medical Illness (SMI) in patients referred to adult psychiatry by emergency physicians, as well as to determine admission rates for SMI soon after discharge from an inpatient psychiatry admission.

ELIGIBILITY:
Inclusion Criteria:

* All patients greater than or equal to 18 years of age presenting to London Health Sciences Centre, Victoria Hospital emergency department between October 1, 2014 - July 31, 2015 who were referred to adult psychiatry by the emergency physician.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients greater than or equal to 18 years of age presenting to London Health Sciences Centre, Victoria Hospital emergency department between October 1, 2014 - July 31, 2015 who were referred to adult psychiatry by the emergency physician
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
number of referrals to medical/surgical consult services within 14 days of psychiatric referral | 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- Victoria site, London Health Sciences Centre, London, Ontario, Canada